CLINICAL TRIAL: NCT01668667
Title: Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose, Parallel-Group Study to Compare the Efficacy, Tolerability, and Safety of 3 Doses of Gabapentin Enacarbil (GSK1838262) With Placebo in Treatment of Moderate-to-Severe Primary RLS
Brief Title: Gabapentin Enacarbil (GSK1838262) Adult Restless Leg Syndrome (RLS) Post Marketing Commitment Study
Acronym: CONCORD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114025
Record Dates: First submitted 2012-06-14; First posted 2012-08-20 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Restless Legs Syndrome
Keywords: gabapentin enacarbil; Horizant
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin; 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK1838262 600 mg (Active Comparator): Once-daily dose with food in the evening at approximately 5 PM
  Interventions: Drug: GSK1838262 600 mg
- GSK1838262 450 mg (Active Comparator): Once-daily dose with food in the evening at approximately 5 PM
  Interventions: Drug: GSK1838262 450 mg
- GSK1838262 300 mg (Active Comparator): Once-daily dose with food in the evening at approximately 5 PM
  Interventions: Drug: GSK1838262 300 mg
- GSK1838262 placebo match (Placebo Comparator): Once-daily dose with food in the evening at approximately 5 PM
  Interventions: Drug: GSK1838262 Placebo match

INTERVENTIONS:
Drug: GSK1838262 600 mg — Drug: GSK1838262 600 mg/day Comparison of 3 doses
  Other Names: Horizant; gabapentin enacarbil GEn; XP13512
  Arms: GSK1838262 600 mg
Drug: GSK1838262 450 mg — Drug: GSK1838262 450 mg/day Comparison of 3 doses
  Other Names: Horizant; gabapentin enacarbil GEn; XP13512
  Arms: GSK1838262 450 mg
Drug: GSK1838262 300 mg — Drug: GSK1838262 300 mg/day Comparison of 3 doses
  Other Names: Horizant; gabapentin enacarbil GEn; XP13512
  Arms: GSK1838262 300 mg
Drug: GSK1838262 Placebo match — Drug; GSK1838262 placebo to match 600 mg, 450 mg, 300 mg doses
  Arms: GSK1838262 placebo match

SUMMARY:
Gabapentin enacarbil (GEn; GSK1838262; HORIZANT), at a dose of 600 mg/day, is currently approved in the United States for the treatment of adults with moderate-to-severe primary Restless Legs Syndrome (RLS). The aim of this study is to compare the efficacy, tolerability, and safety of GEn at lower doses (450 and 300 mg/day) as well as the already approved dose of 600 mg/day versus placebo for the treatment of subjects with moderate to severe primary RLS. This study is being conducted as a post-marketing commitment (PMC) as a condition of the approval of HORIZANT tablets (NDA 022399).

DETAILED DESCRIPTION:
This is a Phase IV randomized, double-blind, placebo-controlled, fixed-dose, parallel group study to assess the efficacy, tolerability, and safety of 3 doses of GEn (600, 450, and 300 mg/day) compared with placebo in the treatment of subjects with moderate-to-severe primary RLS.

The study will include 9 visits over approximately 14 weeks for eligible subjects including a 1-week Screening Period, a 12-week Treatment Period, and a 1 week Follow up Period. Screening will occur within 1 week of the first scheduled dose of study medication. The total duration of the study, from the first subject enrolled to the last subject completed will be approximately 2 years.

Eligible subjects (at least 18 years of age) must have:

* a diagnosis of RLS according to the IRLSSG Diagnostic Criteria
* a history of RLS symptoms for at least 15 nights in the prior month or, if on treatment, this frequency of symptoms before treatment was started
* documented RLS symptoms for at least 4 of the 7 consecutive evenings/nights during the Screening Period, and a total RLS severity score of at least 15 on the International Restless Legs Syndrome (IRLS) Rating Scale at the screening and baseline visits

Approximately 498 subjects will be enrolled, randomly assigned to treatment groups, and receive study medication once daily for 12 weeks. Subjects will be randomly assigned to receive 1 of the 4 following treatment groups in a ratio of 1:1:1:1:

* GEn 600 mg/day
* GEn 450 mg/day
* GEn 300 mg/day
* Matching placebo

Subjects will be instructed to take their study medication once daily with food in the evening at approximately 5 PM. Each tablet must be swallowed whole and not divided, crushed, or chewed.

Each subject, regardless of treatment assignment, will take 3 tablets of study medication (1 tablet from Bottle A, 1 tablet from Bottle B, and 1 tablet from Bottle C) once daily continuing through the end of the Treatment Period (Week 12). Subjects will return to the study site for a follow-up visit (Visit 9, Week 13) approximately 1 week after the last dose of study medication.

Each subject's participation in the study will be approximately 14 weeks unless they withdraw early from the study. For subjects who complete the study, Visit 9 (which can occur between Day 86 and 92) will be considered their end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older
* History of RLS symptoms for at least 15 nights/month
* Documented RLS symptoms, using the 7-day RLS Symptom Record, for at least 4 of the 7 consecutive evenings/nights during the night
* Total RLS severity score of 15 or greater on the International RLS (IRLS) Rating Scale at Visit 1 and at Visit 2
* Discontinuation of dopamine agonists and/or gabapentin , or other treatments for RLS (e.g. opioids, benzodiazepines) at least 2 weeks prior to Baseline
* If taking any prescription medication, therapy must have been stabilized for at least 3 months prior to Screening with no anticipated changes for the duration of the study
* Female subjects are eligible if of non-childbearing potential or not lactating, has a negative pregnancy, and agrees to use a highly effective method for avoiding pregnancy
* Body mass index of 34 or below
* Estimated creatinine clearance of ≥60 mL/min
* Provides written consent in accordance with all applicable regulatory requirements

Exclusion Criteria:

* History of a sleep disorder that may affect the assessment of RLS
* History of RLS symptom augmentation or end-of-dose rebound with previous dopamine agonist treatment
* Neurologic disease or movement disorder
* Other medical conditions or drug therapy that could affect RLS efficacy assessments or may present a safety concern
* Have clinically significant or unstable medical conditions
* Have active suicidal plan/intent or has had active suicidal thoughts in the past 6 months; has a history of suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (40):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Started | 126 | 125 | 125 | 125
Completed | 95 | 99 | 94 | 102
Not Completed | 31 | 26 | 31 | 23
Not completed — Adverse Event | 3 | 6 | 4 | 4
Not completed — Lack of Efficacy | 3 | 2 | 2 | 3
Not completed — Protocol Violation | 6 | 10 | 12 | 5
Not completed — Lost to Follow-up | 9 | 4 | 7 | 6
Not completed — Physician Decision | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Population: mITT (modified intent to treat) Population: The mITT population will include all randomly assigned subjects who received at least 1 dose (or any portion of a dose) of study medication as defined above for the Safety population, have a baseline IRLS Rating Scale total score, and have at least 1 on-treatment IRLS Rating Scale total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match | Total
Number analyzed (Participants) | 119 | 112 | 111 | 117 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.92) | 52.1 (12.22) | 52.0 (14.51) | 52.1 (13.01) | 51.3 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 69 | 71 | 64 | 277
  Male | 46 | 43 | 40 | 53 | 182
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 6 | 14 | 12 | 8 | 40
  American Indian or Alaskan Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 112 | 97 | 95 | 109 | 413
  White & African American/African Heritage | 1 | 0 | 0 | 0 | 1
  White & Asian | 0 | 0 | 1 | 0 | 1
  Unknown or not Reported | 0 | 0 | 2 | 0 | 2
IRLS Rating Scale Total Score, Continuous [Mean (Standard Deviation); unit: units on a scale] — International Restless Legs Syndrome Rating Scale: Very severe=31-40, Severe=21-30, Moderate=11-20, Mild=1-10, None=0.
  units on a scale | 23.4 (5.61) | 24.0 (5.23) | 23.7 (5.25) | 23.5 (5.34) | 23.6 (5.35)

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to the End of Treatment in the International Restless Legs Syndrome (IRLS) Rating Scale Score
Description: International Restless Legs Syndrome Rating Scale: Very severe=31-40, Severe=21-30, Moderate=11-20, Mild=1-10, None=0.
  Change from Baseline = LOCF value at current visit - value at Baseline (the last nonmissing assessment before the first dose of study medication). A negative treatment difference indicates a benefit relative to placebo.
  The change from baseline data is analyzed using an ANCOVA model with treatment and pooled site as the main effects and the baseline IRLS Rating Scale total score as a covariate.
Time Frame: Baseline, 12 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Number analyzed (Participants) | 119 | 112 | 111 | 117
units on a scale | -12.50 (0.745) | -12.54 (0.764) | -11.48 (0.767) | -9.93 (0.753)
Statistical Analysis 1: Comparison: GSK1838262 600 mg vs GSK1838262 Placebo Match; The null hypothesis for this study is that there is no difference between GEn and placebo in the change from Baseline to the end of treatment in the IRLS Rating Scale total score. All comparisons will be made at the two-sided 0.05 level of significance; Test type: Superiority or Other; p = 0.014, ANCOVA; No adjustment for multiplicity will be made for these analyses; Adjusted mean difference = -2.57, 95% CI 2-sided [-4.62 to -0.52], Standard Error of Mean 0.745 — The change from baseline data is analyzed using an ANCOVA model with treatment and pooled site as the main effects and the baseline IRLS Rating Scale total score as a covariate
Statistical Analysis 2: Comparison: GSK1838262 450 mg vs GSK1838262 Placebo Match; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, ANCOVA; No adjustment for multiplicity will be made for these analyses; Adjusted mean difference = -2.61, 95% CI 2-sided [-4.68 to -0.54], Standard Error of Mean 0.764 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GSK1838262 300 mg vs GSK1838262 Placebo Match; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.144, ANCOVA; No adjustment for multiplicity will be made for these analyses; Adjusted mean difference = -1.55, 95% CI 2-sided [-3.63 to 0.53], Standard Error of Mean 0.767 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: The Proportion of Subjects at the End of Treatment Who Are Responders With Either "Much Improved" or "Very Much Improved" on the Investigator-rated Clinical Global Impression of Improvement (CGI-I)
Description: Clinical Global Impression - Improvement Scale (CGI-I): 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), on the scale. Higher score = more affected. Number of subjects responding to treatment at Week 12 with respect to dose level. CGI-I Responders = subjects who reported CGI-I scores of very much improved or much improved.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Number analyzed (Participants) | 119 | 112 | 111 | 117
percentage of participants | 67 | 67 | 68 | 50
Statistical Analysis 1: Comparison: GSK1838262 600 mg vs GSK1838262 Placebo Match; The null hypothesis for this study is that there is no difference between GEn and placebo in the proportion of subjects who are responders with "much improved" or "very much improved" on the investigator-rated CGI-I at the end of treatment; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.30 to 3.95] — The analysis method used was logistic regression with terms of pooled site and treatment
Statistical Analysis 2: Comparison: GSK1838262 450 mg vs GSK1838262 Placebo Match; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.23 to 3.77] — The analysis method used was logistic regression with terms of pooled site and treatment
Statistical Analysis 3: Comparison: GSK1838262 300 mg vs GSK1838262 Placebo Match; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.27 to 3.94] — The analysis method used was logistic regression with terms of pooled site and treatment

3. Secondary Outcome: The Dose-response Relationship of Change From Baseline in IRLS Rating Scale Total Score at End of Treatment
Description: International Restless Legs Syndrome Rating Scale: Very severe=31-40, Severe=21-30, Moderate=11-20, Mild=1-10, None=0.
  This model only includes treatment in the model. Least squares mean is used for analysis.
Time Frame: Baseline, 12 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Number analyzed (Participants) | 119 | 112 | 111 | 117
units on a scale | -12.1 (0.80) | -12.7 (0.82) | -11.3 (0.83) | -9.8 (0.80)
Statistical Analysis 1: Comparison: GSK1838262 600 mg vs GSK1838262 450 mg vs GSK1838262 300 mg; For the mean change from Baseline for IRLS Rating Scale total score at the EOT, the linear contrast test based on an analysis of variance with treatment effect was used to detect linear dose-response trends across increasing levels of GEn dosage; Test type: Superiority or Other; p = 0.022, ANOVA
Statistical Analysis 2: Comparison: GSK1838262 600 mg vs GSK1838262 450 mg vs GSK1838262 300 mg; Overall treatment effect; Test type: Superiority or Other; p = 0.072, ANOVA

4. Secondary Outcome: The Dose-response Relationship for Investigator-rated CGI-I Scale at End of Treatment
Time Frame: 12 Weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Number analyzed (Participants) | 119 | 112 | 111 | 117
percentage of participants
  Responder | 67 | 67 | 68 | 50
  Non-Responder | 33 | 33 | 32 | 50
Statistical Analysis 1: Comparison: GSK1838262 600 mg vs GSK1838262 450 mg vs GSK1838262 300 mg; Test type: Superiority or Other; p = 0.012, Cochran-Armitage trend test — A significant p-value will indicate a nonzero linear effect across increasing levels of GEn dosage

ADVERSE EVENTS:
Time Frame: AEs are collected from the start of study medication and until the follow-up contact. SAEs are collected over the same time period as AEs. SAEs related to study participation are recorded from the time of consenting up to & including any follow-up contact
Description: All safety summaries were based on Safety Population, which was defined as all subjects who received at least 1 dose or any portion of a dose of study medication.
Groups:
- GSK1838262 Placebo Match: Once-daily dose with food in the evening at approximately 5 PMmatching placebo.
Arm/Group | GSK1838262 600 mg | GSK1838262 450 mg | GSK1838262 300 mg | GSK1838262 Placebo Match
Serious Adverse Events (participants affected / at risk) | 1/122 | 0/123 | 2/121 | 1/121
Other Adverse Events (participants affected / at risk) | 55/122 | 56/123 | 33/121 | 46/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1838262 600 mg (N=122) | GSK1838262 450 mg (N=123) | GSK1838262 300 mg (N=121) | GSK1838262 Placebo Match (N=121)
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Unrelated treatment emergent SAE
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 — Unrelated treatment emergent SAE
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 — Unrelated treatment emergent SAE
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Unrelated treatment emergent SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1838262 600 mg (N=122) | GSK1838262 450 mg (N=123) | GSK1838262 300 mg (N=121) | GSK1838262 Placebo Match (N=121)
Somnolence (Nervous system disorders) | 13 | 20 | 12 | 8 — Treatment Emergent AE
Headache (Nervous system disorders) | 11 | 9 | 10 | 12 — Treatment Emergent AE
Dizziness (Nervous system disorders) | 15 | 8 | 5 | 5 — Treatment Emergent AE
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 3 | 7 — Treatment Emergent AE
Nausea (Gastrointestinal disorders) | 5 | 4 | 3 | 7 — Treatment Emergent AE
Fatigue (General disorders) | 5 | 5 | 0 | 7 — Treatment Emergent AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.